CLINICAL TRIAL: NCT02859714
Title: Detection of Colorectal Adenomas in Côte-d'Or: Impact of Organized Screening on Socio-geographic Disparities
Brief Title: Detection of Colorectal Adenomas in Côte-d'Or
Acronym: DACCOR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: COTTET PARI 2015
Record Dates: First submitted 2016-08-01; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- colorectal adenoma
  Interventions: Other: screening data

INTERVENTIONS:
Other: screening data

SUMMARY:
Previous studies have shown geographic disparities in the detection of colorectal adenomas in Côte-d'Or, with an impact of the distance from the general practitioner and an ecological deprivation index (EDI). On the other hand, the extremely low detection rates for these lesions in everyday practice before the implementation of organized screening for colorectal cancer in the Côte-d'Or were shown. One of the aims of this screening is to reduce socio-geographic inequalities in access to care and prevention. Yet, participation in screening also varies depending on the socio-economic level. In this context, the Côte-d'Or Polyps Registry, the only body to have data for the pre-screening period (before 2003), will make it possible to determine whether the implementation of organized screening led to the elimination of socio-geographic disparities concerning the detection of adenomas.

ELIGIBILITY:
Inclusion Criteria:

* The study population will include all patients residing in Côte d'Or with a first colorectal adenoma (including in situ carcinomas) diagnosed between 01/01/1997 and 31/12/2008

Exclusion Criteria:

* Absence of address
* history (or suspected history) of previously resected adenoma
* personal history of colorectal cancer or colorectal cancer discovered in the year following resection of the adenoma (because the cancer was probably not seen at the initial colonoscopy)
* familial polyposis or known HNPCC
* chronic inflammatory bowel disease

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients residing in Côte d'Or with a first colorectal adenoma (including in situ carcinomas) diagnosed between 01/01/1997 and 31/12/2008.
Sampling Method: Non-Probability Sample
Enrollment: 11600 (Estimated)
Dates: Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Detection rates for colorectal adenomas | through the study completion up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France